CLINICAL TRIAL: NCT04292275
Title: A Randomized, Open-Label, Standard-of-Care-Controlled, Multicenter Study to Evaluate Digital Health Data Use in Managing Guideline-Directed Heart Failure Therapy
Brief Title: Heart Failure Study to Evaluate Vital Signs and Overcome Low Use of Guideline-Directed Therapy by Remote Monitoring
Acronym: HF-eVOLUTION
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed prematurely due to enrollment challenges exacerbated by COVID-19.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20180096
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: Digital health; Remote monitoring; Wearable device
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Health Tools + Standard of Care (Experimental)
  Interventions: Device: Biobeat Wrist Watch; Other: Standard of Care
- Standard of Care (Other)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Biobeat Wrist Watch — Standard of care procedures and therapies for managing heart failure will be carried out according to each investigator's standard procedures. In addition, participants will be provided with a Biobeat wrist watch for continuous measurement and reporting of blood pressure data and with a smartphone to report weight.
  Arms: Digital Health Tools + Standard of Care
Other: Standard of Care — Standard of care procedures and therapies for managing heart failure will be carried out according to each investigator's standard procedures.

SUMMARY:
A study evaluating the impact of remotely collected data, measured using digital technologies, on the use of guideline-recommended heart failure therapy in adult participants with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic heart failure.
* Ejection fraction equal to or below 40%.
* New York Heart Association (NYHA) class II to class III.
* Enrollment during or within 30 days after a hospitalization, emergency department, or urgent, unscheduled clinic/office visit with primary diagnosis of heart failure.

Exclusion Criteria:

* Has received a major organ transplant (e.g., lung, liver, heart, bone marrow, kidney).
* Currently in an investigational device or drug study.
* Unwilling or unable to wear a digital wrist watch device for measuring blood pressure and other parameters during waking hours.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Time to Change or Decision That Heart Failure Therapy is Optimal | Randomization to 6 months
  Area under the curve (AUC) will be calculated for a daily dose-related medication score for beta-blocker, angiotensin-converting enzyme inhibitor/angiotensin II receptor blocker/angiotensin neprilysin inhibitor, and aldosterone antagonist therapy.

SECONDARY OUTCOMES:
Time to change or decision that heart failure therapy is optimal | Baseline to 6 months
  Area under the curve (AUC) will be calculated for a daily dose-related medication score for beta-blocker, angiotensin-converting enzyme inhibitor/angiotensin II receptor blocker/angiotensin neprilysin inhibitor, and aldosterone antagonist therapy, time to change or decision that dose is optimal.
Numerical Health Information Technology Usability Evaluation Scale for Healthcare Provider Scores (Health-ITUES-HCP) | Week 24
  Health-ITUES-HCP will be used to assess the healthcare provider's experience with the digital health tool(s) and data presentation. The scale consists of 36 items. A higher score indicated higher perceived usability of the technology.
Numerical Health Information Technology Usability Evaluation Scale for Participants (Health-ITUES-Subject) Scores | Week 24
  Health-ITUES-Subject will be used to assess the participant's experience with the digital health tool(s). The scale consists of 36 items. A higher score indicated higher perceived usability of the technology.
Change in Numerical Rating of Subject Satisfaction with Heart Failure Therapy | Baseline and Week 24
  Participants will complete a subject satisfaction survey (5 point Likert scale format) ranging from very satisfied to very dissatisfied.
Change from Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ-23) Scores | Baseline and Week 24
  The KCCQ-23 is a 23-item questionnaire to measure the participant's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life. All items are measured on a Likert scale with 5-7 response options. Scores for each item are standardized to range from 0 to 100 with higher scores indicating better health status, fewer symptoms, and greater disease-specific health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (8):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Cardiology Associates of Fairfield County, PC, Stamford, Connecticut
  - MercyOne Northeast Iowa Family Medicine and Residency, Waterloo, Iowa
  - Virtua Health Inc., Voorhees Township, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Diagnostic Cardiology Group, Chattanooga, Tennessee
  - Tennessee Center for Clinical Trials, a division of Cardiology and Vascular Associates PLLC, Tullahoma, Tennessee
  - Inova Heart and Vascular Institute, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com